CLINICAL TRIAL: NCT01264991
Title: The Benefit of Arthroscopic Partial Meniscectomy in Middle-Aged Patients - A Double-Blinded Randomized Placebo (Sham) Controlled Multi-Centre Trial
Brief Title: The Benefit of Arthroscopic Partial Meniscectomy in Middle-Aged Patients
Acronym: SLAMSHAM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment stalled. Study terminated before inclusion of sufficient number of participants included
Sponsor: Slagelse Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Kristoffer Hare, MD, Slagelse Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SJ-183
Record Dates: First submitted 2010-12-21; First posted 2010-12-22 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Degenerative Meniscus Tear
Keywords: Sham; Meniscus tear; Meniscectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- APM group (Experimental)
  Interventions: Procedure: Arthroscopic partial meniscectomy
- Sham group (Placebo Comparator)
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Procedure: Arthroscopic partial meniscectomy — The arthroscopic partial meniscectomy will be performed on an outpatient basis by experienced surgeons at a level of at least attending physicians or at the last year of residency. All arthroscopies will be performed in general anaesthesia combined with local anaesthesia. After general anaesthesia is induced, the knee will be examined for stability. Thereafter two standard portals on the lateral and medial side of the ligamentum patella will be created but no outflow cannula inserted. An arthroscope will be used with a pressure-controlled irrigation system. Tourniquet use will be according to surgeon preference. The strategy for the meniscectomy will be to preserve as much tissue as possible. A standard operation protocol will be used to document possible findings in cartilage, ligaments, synovium and the medial and lateral meniscus. Meniscus lesions and type of will be registered and changes in the articular cartilage will be classified according to the ICRS classification
  Arms: APM group
Procedure: Sham procedure — The placebo procedure will be performed under the same conditions as above. The patient will be fully sedated in general anaesthesia. As above, the stability of the knee will be examined. Local anaesthetic will be applied as above and 2 skin incisions will be made at the same location and the same size as above. Then the knee will be manipulated as if a real arthroscopy were being done, the spillage of water and all the other equipment needed for an arthroscopy will be used and manipulated. No instruments will enter the portals for arthroscopy to avoid the possibility of osteochondral lesions and unwanted interventions by the surgeon.
  Arms: Sham group

SUMMARY:
BACKGROUND Osteoarthritis (OA) is the most common form of arthritis and the knee is one of the most affected joints. The meniscus plays an important role in the development of knee OA. It is unclear whether a degenerative meniscus tear is a risk factor in developing knee OA or a sign of the disease. The standard treatment for a degenerative meniscus tear is an arthroscopic partial meniscectomy (APM). There is strong evidence that this puts the knee at high risk of later developing OA. Earlier studies have shown a significant placebo effect from surgical procedures, in general, and an arthroscopic knee procedure, in particular.

PURPOSE The overall purpose of this study is to gather information that might lead to a reduction in the development of OA in middle-aged patients. The investigators hypothesise that the benefit from an arthroscopic partial meniscectomy is due to the placebo effect measured on self-reported outcomes, and that the meniscectomy contributes to the development of knee OA as seen on radiography.

METHODS The investigators will include 100 patients aged from 35 to 55 years with an MRI-confirmed medial meniscus tear and without knee OA (excluding patients with Grade 3 or 4 knee OA on the Kellgren-Lawrence classification). Participants will be randomised to either a standard APM procedure or a sham procedure and both groups will receive standard post-operative care. The primary outcomes will be a self-reported questionnaire, the KOOS score, and a functionality test after 3 and 24 months.

DETAILED DESCRIPTION:
BACKGROUND Osteoarthritis (OA) is the most common form of arthritis and affects 4.5 % of the Danish population. The knee is one of the most affected joints and 45 % of all OA-related hospital contacts are related to the knee. OA has a long 'pre-clinical' phase with joint changes without symptoms. Then comes a symptomatic phase with pain and functional limitations. This is sometimes accompanied by structural changes visible on plain X-ray examination and other pathological changes like focal areas of damage to the articular cartilage, centered on load-bearing areas. After this, new bone formation at the joint margins (osteophytosis) develops along with changes in the subchondral bone, variable degrees of mild synovitis, and thickening of the joint capsule.

The meniscus plays an important role in the development of osteoarthritis. Meniscus tears can be both a risk factor for knee OA as well as a sign of disease . Both meniscus injury and a meniscectomy contribute to the development of knee OA. The surgical removal of the damaged parts of a meniscus tear puts the knee at high risk of later developing OA . Surgical resection also leads to increased joint cartilage contact stress through altered load transmission, decreased shock absorption, and decreased joint stability .

The current standard treatment for a degenerative meniscus tear is arthroscopic partial meniscectomy (APM). Arthroscopic surgery is one of the most frequent orthopaedic procedures with approximately 10,000 APM procedures being done per year in Denmark .

The benefit from an APM procedure is, however, uncertain and needs to be further investigated. As mentioned above, it significantly increases the risk of developing knee OA. The investigators also know that a significant placebo effect is present in arthroscopic knee surgery including the APM procedure . It has furthermore been shown that patients with a degenerative meniscus tear can recover without surgery and by exercise alone , . The recovery period after an APM procedure is also much longer than most surgeons realize, with disability still evident after 3 months.

The investigators need to investigate the placebo effect in younger patients with a degenerative meniscus tear but without knee OA by implementing additional well-designed, randomized, placebo controlled trials to reveal the true effects of the APM procedure on a short-and long-term basis.

The benefit, on a short- and long term basis of APM are firstly described in non-controlled studies from the 1980-90's. , , when arthroscopic surgery were gaining entry. But poorly designed studies (retrospective, use of non-validated outcome scores, small patient populations) and the lack of randomised studies has not shown the true effect of the APM procedure. A Cochrane review from 2000(withdrawn due to age) concludes:"…lack of randomised trials means that no conclusions can be drawn on the issue of surgical versus non-surgical treatment of meniscus injuries". This is up to this point no studies that shows a positive benefit from APM compared to other treatment modalities. Those studies that exist beyond this point (Moseley 2003, Herrlin 2007, Kirkley 2008) has not shown APM to be better than other treatments (placebo, physiotherapy, medication or exercise). The patients though in these studies were of older age (mean 52 to 62 years) and had already developed symptomatic knee OA. There is but one study of recent age of non-surgical treatment of meniscus tears on younger patients (n32) which recommends an initial course of non-operative treatment. The investigators wish to examine whether the same conditions which applies to the elder patients with knee OA also apply to the younger patients without knee OA.

A mathematical model has been proposed to identify which patients will receive a benefit or not from the APM procedure because, according to the author, an RCT would be controversial with reluctance and lack of equipoise from both surgeons and patients . Meanwhile several editorials suggest that the use of sham procedures should play a larger role in orthopaedic surgery research , , . Furthermore, a recent study of vertebroplasty showed the need for placebo-controlled surgical trials to avoid widespread adoption of new unnecessary interventions in routine care.

ETHICAL CONSIDERATIONS The first thought that comes to many people when introduced to this protocol is: "Is it ethical to perform placebo-controlled RCTs of surgery? However, the initial precept in medicine is "First, do no harm". For example, one cannot imagine a new pharmaceutical product to be marketed without its being compared with a placebo or at least to a similar drug. The investigators assume this process has been undertaken, in spite of the likely adverse effects from any drug.

An equally valid question is, 'Is it ethical not to perform placebo-controlled RCTs within orthopaedics and instead, potentially perform under-researched operations which may not benefit the patient, or actually, do harm?' As mentioned earlier, a recent study of vertebroplasty has effectively shown how a placebo-controlled surgical trial can evaluate a given procedure that has been adopted widely despite an absence of robust evidence.

There are three reasons to perform another placebo-controlled arthroscopy study apart from Moseley's (2003). First, this study will focus on younger patients, second these patients are yet to develop knee OA but are at risk of doing so, and third, a replication study is required to make Moseley's evidence convincing.

A multistep process has been proposed to ensure that sham-controlled surgical trials are performed in an ethical manner :

1. There is scepticism regarding the therapeutic merits of a particular surgical treatment
2. There are disagreements about the perceived benefits of a particular procedure compared with the placebo.
3. Benefits might be due to the "experience of surgery" and the postoperative care regimen.
4. Risks are reduced as far as possible in the sham surgery arm without compromising trial design.
5. There is a lack of a superior alternative therapy.

   Using the model above, our study would have the following basis:

   Ad 1) The APM procedure is controversial. The investigators know that it will lead to knee OA.

   Substantial disability has been shown after the APM procedure. Ad 2) Earlier studies have shown a significant placebo effect in arthroscopic surgery for knee OA. Other studies have shown no difference in surgical or non-surgical treatment of degenerative meniscus tears.

   Ad 3) As has been shown patients can recover even from degenerative meniscus tears with mechanical symptoms suggesting that the benefit from a surgical intervention can be due to the "experience of surgery" and the usual postoperative regime.

   Ad 4) The risk is minimized to a skin incision and general anaesthesia. The overall complication risk from a knee arthroscopy is 0.5% . Only relatively healthy patients eligible for outpatient surgery are included to avoid an increased risk during the anaesthesia.

   Ad 5) Alternative therapies are medical treatment and/or exercise, but the literature has not yet shown superiority over the APM procedure.

   PURPOSE The overall purpose of this study is to test whether the benefit from an APM in patients aged 35-55 with knee pain and a meniscus lesion, is due to the surgery or to the placebo effect. Demonstration of no additional benefit from this surgery may reduce the development of surgically-related osteoarthritis in middle-aged patients.

   The investigators hypothesize that the benefit from an arthroscopic partial meniscectomy measured on self-reported outcomes is due to the placebo effect, and that meniscectomy contributes to the development of knee osteoarthritis seen on radiography.

   PROJECT DESIGN The study is designed as a prospective double-blinded randomized placebo-controlled multicentre trial. Patients will be randomized to receive either an APM or placebo (sham) procedure. The patients will furthermore be stratified into those with and without mechanical symptoms.

   Patients referred from general practitioners will be screened initially. If eligible, written information about the study including a 10 minute video will be given to the patients to view at home. They will also be handed the questionnaires to fill out at home. At the second contact the patients will receive an MRI scan of the affected knee and perform a physical function test. After this the patients are informed of the MR findings. If MRI confirms medial meniscus lesion the patient will be included in the study and signed up for surgery.

   At 3 months, the patients will be called in for a follow-up which will include a physical function test, an objective examination and a request to fill out a questionnaire. At 2 years, a new follow-up will take place under the same conditions.

   Postoperative regime All patients in both intervention groups will be given a folder including an exercise program for postoperative patients after knee arthroscopy. The folder gives a presentation of 7 different non-weight bearing exercises (for the first week after surgery) and a further 3 weight bearing exercises thereafter. The exercises are for the patients to carry out at home. The patients are also recommended to start unloaded cycling, swimming or walking after 1 week and after 2-3 weeks the patients are recommended jogging or loaded cycling.

   Considerations regarding anaesthesia:

   In this study all patients will be given general anaesthesia. Considerations about minimizing the patient risk in the placebo group have been either to induce deep sedation or general anaesthesia. In Moseley's study the patients in the placebo group were only sedated to minimize the risk. This is a lot like in an endoscopy setting, where the use of deep sedation with Propofol has been in wider use. In that setting the goal is to complete the procedure without the need for an anesthesiologist thus reducing the costs of the procedure. There are still complications associated with deep sedation . No study exists which compares the complication risk of general anaesthesia with deep sedation, but the incidence of complications in deep sedation in an endoscopy setting compared with general anaesthesia in an arthroscopy setting seems the same . In this study there is no account to the cost of the procedure only to the risk of the patient. Therefore general anaesthesia with superior airway control versus deep sedation and also with no risk of compromising the study design has been chosen.

   A surgical checklist has previously shown to decrease mortality and will be used for all patients in this study to insure safety. An attending anesthesiologist will be responsible for the anesthesia either directly or as a supervisor. All patients will be fully sedated with Ultiva/Propofol and a larynx mask will be applied. The overall risk of death by anesthesia is 1:250.00 in healthy patients and in Denmark 3 deaths per year have been reported due to anesthesia There are 3 reasons why regional anesthesia has not been chosen. First, blinding the patient will be much more difficult if he is awake, due to the manipulation of the knee, the time perspective and none the less the "acting" from the operational staff which is required. Second, no outpatient clinic in Hospital South, Region Zealand offers regional anesthesia at this moment. Third, study design may be compromised by having a non-homogenous group of patients receiving different kind of anesthesia. Studies have shown that though regional anesthesia is a preferable option in outpatient arthroscopic surgery it has not been shown to be less in healthy individuals .

   Patient characteristics and baseline At baseline, a registration of gender, weight, height, working status and level of education will be collected.

   After surgery the patients will be asked which procedure they think they have been through. Likewise patients will be asked of their expectations to the surgical procedure and afterwards if these expectations were fulfilled.

   A questionnaire of patient self-efficacy modified after the Danish Arthritis Self-Efficacy Score will be included.

   Objective and subjective mechanical findings (decreased range of motion, clicks, locking) will be registered.

   All patients will receive:
   1. A clinical examination (joint line tenderness, range of motion, swelling, mechanical findings, McMurray test)
   2. Weight-bearing x-rays of both knees
   3. MRI of the affected knee
   4. A functionality test
   5. Questionnaires (see "Outcome")

   RADIOLOGY All MRI's will be conducted at the same location and reviewed by the same radiologist. A meniscus tear, maceration, and/or destruction are graded according to the Whole-Organ MRI Score (WORMS) method (28). The anterior horn, body segment, and the posterior horn of the medial and lateral menisci were graded separately on a scale of 0-4, where 0 = intact, 1 = minor radial or parrot-beak tear, 2 = non-displaced tear (breaking 2 or more surfaces), 3 = displaced tear or partial maceration or destruction, and 4 = complete maceration or destruction. The readers regarded an increased intra-meniscus signal (often a linear signal within the meniscus) as a meniscus tear when it communicated with the inferior or superior margin of the meniscus on at least 2 slices.

   X-ray of both knees with the patient standing will be taken at a fixed flexion angle using the Synarflexer. Classification of osteoarthrosis will be according to Kellgren-Lawrence classification:

   Grade 0 No radiographic findings of osteoarthritis Grade 1 Minute osteophytes of doubtful clinical significance Grade 2 Definite osteophytes with unimpaired joint space Grade 3 Definite osteophytes with moderate joint space narrowing Grade 4 Definite osteophytes with severe joint space narrowing and subchondral sclerosis

   All patients will be asked for reasons to participate in the study, or to decline, and in either case they will be asked which material was helpful in making that decision (written information, the video or other) and other reason for their choice (e.g. wanting to contribute to the research, not wanting a sham procedure etc.).

   PHYSICAL FUNCTION TEST Single leg hop test The investigators will include a single leg hop test, the one-leg hop . Subjects will perform 2 practice trials and then two test trials on each leg. The best of the two test trials will be used. Symmetry indices will be calculated for the one-leg hop test as (injured side/uninjured side) x 100.

   Knee-bending test The investigators will also include maximum number of knee-bends performed in 30 seconds as a third test for physical function. This test has been used on similar patient groups in other studies , , and has been found to be a reliable test .

   Muscle strength test A handheld dynamometer (Powertrack Commander) will be used to evaluate the quadriceps muscle performance by measuring the knee-extension strength. Isometric muscle testing is commonly used in the literature and the reliability for the isometric muscle tests with a hand held dynamometer have previously been reported to be satisfactory .

   Prior to the muscle and functional tests, subjects will warm up on a stationary bicycle for approximately 10 minutes. The responsible test facilitator will be blinded to which knee is affected by led the patient wear a neoprene sleeve over both knees. In order to decide which leg is tested first the patient will be randomized at each visit to avoid bias from the effect of learning.

   ADVERSE EVENTS

   All complications or adverse events associated with both interventions will be registered; Infection (deep or superficial), deep-vein thrombosis, nerve or vessel injury or compartment syndrome. An adverse event is defined as any unwanted event. A serious adverse event is defined as an event that could lead to:
   1. Death
   2. A threat to life
   3. Hospitalization
   4. Some form of handicap
   5. Congenital defects
   6. A significant medical condition

   Expected adverse events are:

   Superficial infection, Nerve or vessel injury, Deep infection, Compartment syndrome, Deep venous thrombosis, Myocardial infarction, Stroke, Death.

   All adverse events (including those not anticipated in the table above) will be gathered from journal review, from the national database index and from the follow-ups at 3 and 24 months.

   SAMPLE SIZE This is based on a superiority study. A sample size calculation was done using a standard formula. SD,the standard deviation is defined as 15, in order to make this study comparable with other studies using the KOOS score.

   Z, the standard normal distribution with a probability of a Type I (here 0.05) and Type II error (usually between 0.05 and 0.20. Here decided on 0.1 = a power of 90%. D is the clinical importance or relevant difference. In these calculations 10/100 points for the KOOS questionnaire subscales is chosen as a clinical important or relevant difference.

   Based on above forty patients are needed in each group. With an expected drop-out rate of about 20 %, the investigators intend to recruit 50 patients for each group resulting in a total of 100 patients.

   RANDOMIZATION The investigators will use a computer-generated randomization schedule where annotations for treatment according to meniscectomy (A) or placebo (B) will be used. To ensure an equal distribution in the two groups, the investigators will use a block randomization, using blocks of 4 and 6. Participants will be stratified to each treatment center.

   To ensure concealment of the assigned intervention, the surgeon will obtain the sealed envelope containing the participant's assigned intervention after the patient is in the operating suite and has been fully sedated. The envelope will be retrieved from a briefcase located at the actual operating theatre.

   The allocation sequence will be generated by an external co-investigator, the enrollment will be performed by the author and the assignment will be at the operating room when the envelopes will be opened by the surgeon.

   The treating surgeon will have no other role in the trial.

   BLINDING The RCT will be a double-blinded study. All study personnel and participants will be blinded to the intervention except for the surgeons, who do not have any other role in the study and the external statistician who will be presented to the unblinded data.

   STATISTICAL METHOD All subjects assigned to treatment will be included in the efficacy analyses (i.e. intention to treat analysis). Between-group comparisons of the primary end point will be made with the use of a random effects model. 10/100 points for the KOOS questionnaire subscales are chosen as a clinical important or relevant difference, thus a confidence interval excluding differences greater than 10 units between groups is interpreted as indicating the absence of a clinically meaningful difference.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with knee pain for more than 2 months without significant trauma (only the index knee will be included)
2. MRI-confirmed medial meniscus lesion (patients with a medial meniscus lesion AND a lateral lesion will also be included)
3. Age 35-55 years*
4. Eligible for outpatient surgery - ASA score 1-2

Exclusion Criteria:

1. Patients in need of acute surgery e.g. locking knees, high-energy trauma
2. Symptoms associated with other musculoskeletal co-morbidities overriding the symptoms of the knee
3. Grade 3 or 4 knee OA on the Kellgren-Lawrence classification
4. Knee surgery within the last 2 years
5. Obese patients with BMI > 35
6. Patients with ischemic heart disease
7. Patients with diabetic late-complications
8. Patients with thrombophilia
9. Pregnancy
10. Patients unable to speak Danish
11. Patients with drug or alcohol abuse

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2011-02-21 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score - KOOS | 2 year follow-up
  The primary outcome at 2 years follow-up will be a self-reported questionnaire, the Knee injury and Osteoarthritis Outcome Score (KOOS), comprising five different subscales:
  1. pain
  2. other symptoms
  3. activities in daily living (ADL)
  4. function in sport and recreation
  5. knee-related quality of life (QOL) A mean of the 5 subscales will be calculated (KOOS5 = [KOOSpain + KOOSsymptoms + KOOSADL + KOOSsport&rec KOOSQOL] / 5. Range 0 to 100, worst to best)

SECONDARY OUTCOMES:
One-leg jump test | 2 year follow-up
  Subjects will perform 2 practice trials and then two test trials on each leg. The best of the two test trials will be used. Symmetry indices will be calculated for the one-leg hop test as (injured side/uninjured side) x 100
Knee-bending test | 2 year follow-up
  A maximum number of knee-bends performed in 30 seconds as a test for physical function. This test has been used on similar patient groups in other studies and has been found to be a reliable test
Knee extension strength | 2 year follow-up
  A handheld dynamometer (Powertrack Commander) will be used to evaluate the quadriceps muscle performance by measuring the knee-extension strength. Isometric muscle testing is commonly used in the literature and the reliability for the isometric muscle tests with a hand held dynamometer have previously been reported to be satisfactory.
EQ-5D | 2 year follow-up
  The EQ-5D health score will be evaluated at baseline and at 3 and 24 months as a generic measure of health for clinical and economic appraisal. EQ-5D consists of two pages - the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, severe problems.
SF-36 | 2 year follow-up
  The SF-36 Health Survey - Acute (1 week re-call) will be used as a generic measure of patient health status and in differentiating the health benefits produced by the different treatments. This will also be evaluated at baseline and at 3 and 24 months. The SF-36 Is compromised of an 8-scale profile of functional health and well-being scores comparing the relative burden of diseases.
Development of knee osteoarthritis | 5 year follow-up
  A fixed-flexion radiography procedure, with use of SynaFlex, will be implemented to investigate the development of OA on a long-term basis . Incident marginal tibiofemoral osteophyte will be the outcome at a 5-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Roos, Professor, Study Chair — Research Unit of Musculoskeletal Function and Physiotherapy, Institute of Sports Science and Clinical Biomechanics, University of Southern Denmark, Odense; Kristoffer B Hare, MD, Principal Investigator — Dept. of Orthopadeics, Slagelse Hospital, Region Zealand
Locations (2):
- Denmark (2):
  - Næstved Hospital, Næstved, Region Sjælland
  - Slagelse Hospital, Slagelse, Region Sjælland

REFERENCES:
- [Derived] Roos EM, Hare KB, Nielsen SM, Christensen R, Lohmander LS. Better outcome from arthroscopic partial meniscectomy than skin incisions only? A sham-controlled randomised trial in patients aged 35-55 years with knee pain and an MRI-verified meniscal tear. BMJ Open. 2018 Feb 2;8(2):e019461. doi: 10.1136/bmjopen-2017-019461. PMID 29420232
- [Derived] Hare KB, Lohmander LS, Roos EM. The challenge of recruiting patients into a placebo-controlled surgical trial. Trials. 2014 May 13;15:167. doi: 10.1186/1745-6215-15-167. PMID 24884948
- [Derived] Hare KB, Lohmander LS, Christensen R, Roos EM. Arthroscopic partial meniscectomy in middle-aged patients with mild or no knee osteoarthritis: a protocol for a double-blind, randomized sham-controlled multi-centre trial. BMC Musculoskelet Disord. 2013 Feb 25;14:71. doi: 10.1186/1471-2474-14-71. PMID 23442554